CLINICAL TRIAL: NCT02240420
Title: Reaching High Risk Post-partum Women for Nutritional Assessment and Counseling Via a Telephone-based Coaching Program
Brief Title: Diabetes Prevention Among Post-partum Women With History of Gestational Diabetes
Acronym: Star-Mama
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Department of Public Health (Other Government); San Francisco General Hospital (Other); Sonoma Department of Public Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CFDA 10.586
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Gestational Diabetes Mellitus; Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes prevention in the post-partum; Behavior change among Latinas,; Health Coaching, Motivational interviewing techniques
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Hybrid type 1 effectiveness implementation design, focusing on weight loss and behavior change outcomes, as well as engagement and acceptability of the intervention
Oversight: Data Monitoring Committee: No

ARMS (2):
- Life Style counseling (Star-Mama) (Active Comparator): Star-Mama intervention group will receive during 6 months weekly phone calls with queries and narratives about health habits. The participant's answers will be sent to a health coach who will follow up with the participant, and develop a plan with the participant to address her needs.
  Interventions: Behavioral: Life Style Counseling (Star-Mama)
- Educational Resource Support (No Intervention): Participants in the control group of the study will receive a set of educational materials with information about their health and the health of their babies.

INTERVENTIONS:
Behavioral: Life Style Counseling (Star-Mama) — Participants enrolled in the Star-Mama intervention group will receive 1. weekly automated phone calls with prevention-focused queries (e.g., diet, exercise, breastfeeding). 2. If a participant generates a value rated "out of range," a health coach who receives daily electronic downloads of STAR-Mama responses will call the participant to coach her about the specific health issue. Participants also hear recorded narratives related to their "out of range" reply encouraging behavior change. 3. Call-backs enable coaches to engage patients in goals setting/action plans and providing information about community resources
  Other Names: Star-Mama intervention
  Arms: Life Style counseling (Star-Mama)

SUMMARY:
The purpose of the STAR-MAMA intervention is to develop a patient-tailored telephone-base counseling intervention for young Latino women who are at high risk of diabetes. The intervention will focus at the end of pregnancy and the 9 months post-partum period to improve education and behavioral counseling on nutrition and other related health topics .

The following hypotheses will be formally tested:

Compared with controls at 9 months post-partum:

1. Women in the STAR-Moms program will have improved self-reported behavioral outcomes for minutes of physical activity, lower fat diet, and breast-feeding duration (in weeks);
2. Women in the STAR-Moms program will have improved diabetes prevention knowledge;
3. Women in the STAR-Moms program will have increased diabetes-relevant screening rates.

Women in the STAR-MAMA will have lost more weight than women in the control group.

DETAILED DESCRIPTION:
The STAR-MAMA intervention builds on theoretical constructs found in Social Cognitive Theory, Theory of Planned Behavior, and Theories of Social Support found to be effective in weight loss, physical activity and dietary change, based on a recent meta-analysis and other studies. The investigators proposed development of STAR-MAMA will incorporate specific behavior change techniques associated with these theories, including: "self-regulatory" intervention techniques (specific goal setting, prompting self-monitoring, providing feedback on performance, goal review), self-efficacy building intervention techniques (motivational interviewing, using decisional balance and relapse prevention), individual tailoring techniques (information on content and resources), and culturally tailored social support, and which incorporates family needs.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum Latino women (English or Spanish speakers) with history of gestational diabetes.
* 18 years or older

Exclusion Criteria:

* Do not have type 1 or type 2 diabetes.
* Do not have access to phone line or a cellphone to receive weekly calls of health coaching education over the phone.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 181 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-03-10 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Behavior change | 6 month -12 months post-partum
  Women in the intervention arm of the study (Star-Mama) will have behavior changes that lower their risk of developing gestational diabetes in the next pregnancy of type 2 diabetes later in life.

SECONDARY OUTCOMES:
Weight loss | 6-12 months post-partum
  Women in the intervention arm will have weight losses related to improved behaviors on physical activity, healthier nutrition habits and breastfeeding.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret A. Handley, MPH, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Derived] Horwitz MEM, Edwards CV, Athavale P, McCloskey L, Cabral HJ, Benjamin EJ, Handley MA. The STAR-MAMA RCT: Bilingual Mobile Health Coaching for Postpartum Weight Loss. Am J Prev Med. 2023 Oct;65(4):596-607. doi: 10.1016/j.amepre.2023.03.021. Epub 2023 Apr 5. PMID 37028566
- [Derived] Athavale P, Thomas M, Delgadillo-Duenas AT, Leong K, Najmabadi A, Harleman E, Rios C, Quan J, Soria C, Handley MA. Linking High Risk Postpartum Women with a Technology Enabled Health Coaching Program to Reduce Diabetes Risk and Improve Wellbeing: Program Description, Case Studies, and Recommendations for Community Health Coaching Programs. J Diabetes Res. 2016;2016:4353956. doi: 10.1155/2016/4353956. Epub 2016 Oct 26. PMID 27830157
- [Derived] Handley MA, Harleman E, Gonzalez-Mendez E, Stotland NE, Althavale P, Fisher L, Martinez D, Ko J, Sausjord I, Rios C. Applying the COM-B model to creation of an IT-enabled health coaching and resource linkage program for low-income Latina moms with recent gestational diabetes: the STAR MAMA program. Implement Sci. 2016 May 18;11(1):73. doi: 10.1186/s13012-016-0426-2. PMID 27193580